CLINICAL TRIAL: NCT04719442
Title: Translating Efficacious Pediatric Weight Management Interventions Into Rural & Micropolitan Communities
Brief Title: Packaging Building Healthy Families for Community Implementation
Acronym: NECORD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Started record under wrong IRB account. Registered under UNMC, but actually at UNKearney.
Sponsor: University of Nebraska (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 121919-1; 1U18DP006431 (NIH)
Record Dates: First submitted 2020-07-02; First posted 2021-01-22 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Pediatric Obesity
Keywords: Obesity; Type III Hybrid Effectiveness Implementation; Rural
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BHF-LC (Experimental): To test an innovative implementation strategy, four communities will be assigned to pilot test the packaged PWMI and training materials when coupled with a learning collaborative facilitation strategy and sustainability action planning process to support PWMI adoption, implementation, and sustainability (BHF-LC).
  Interventions: Behavioral: Building Healthy Families
- BHF-Program Only (Active Comparator): Four other communities will be assigned to receive the packaged PWMI and training program only.
  Interventions: Behavioral: Building Healthy Families

INTERVENTIONS:
Behavioral: Building Healthy Families — Building Healthy Families (BHF) is a family based obesity treatment program which includes key behavior change strategies including goal setting for both behavior change and weight loss, self-monitoring, rewards/contingency management, role modeling, and stimulus control/ modifying the environment. BHF includes a minimum of 32 contact hours consisting of three main program components: nutrition education, behavior modification, and physical activity. Participants and parents are expected to attend 12 continuous weeks of education (2 hours/session) followed by 12 weeks of relapse prevention refresher courses. Relapse prevention refresher sessions are every three weeks for one hour to re-evaluate goals, discuss rewards/contingency management and changes in stimulus control with seasonal changes and holidays. A final follow-up check-in session is conducted at 12 months for approximately 1 hour.
  Other Names: Building Healthy Families-Program Only

SUMMARY:
There is a large body of literature regarding efficacious intervention strategies for treating childhood obesity. Unfortunately, the degree to which efficacious programs have been packaged for translation in micropolitan and surrounding rural areas is unclear-an important issue when considering the prevalence of obesity is higher in rural areas when compared to urban areas. Epstein's Traffic Light Diet (TLD) is likely the most studied pediatric weight management intervention (PWMI) and has demonstrated efficacy across a wide range of randomized controlled trials in children 6-12 years of age. Building Healthy Families (BHF) is an adaptation of the TLD and has been implemented in a micropolitan city and achieved clinically and statistically significant reductions in child BMI z-score (-0.27±0.22)-a similar magnitude of effect relative to previous efficacy trials. The investigators have created online resources for organizations interested in delivering PWMIs, training modules for related interventions, and participant-facing program materials that could be combined into a 'turn-key' approach for communities interested in reducing childhood obesity to adopt, adapt and sustain it in other micropolitan/rural communities. The primary aim is to collaboratively refine and develop an intervention package for the BHF that includes materials necessary for others to implement the intervention in new metropolitan/rural locations. The second aim is to perform a rigorous, mixed-methods pilot implementation study using an innovative community application process to identify 4 to 8 new communities to pilot test the utility of the packaged PWMI and training materials while determining factors that predict adoption, implementation and sustainability. The investigators will also use a learning collaborative implementation strategy to improve implementation fidelity and local context and facilitation capacity in communities interested in delivering BHF. The third aim is to use the pilot evaluation data and results of the sustainability action plan to refine program and training materials and develop a dissemination plan to move the program to other communities. The approach will use an implementation research explanatory process and outcome model to test hypotheses related to implementation and sustainability, engaging community/ clinical partners in the implementation and sustainability process, and evaluate outcomes at both the individual and organizational level.

DETAILED DESCRIPTION:
Since the early 1980s, a number of efficacious pediatric weight management interventions (PWMI) have been developed to reduce child weight status. Epstein's Traffic Light Diet (TLD) is likely the most studied PWMI and has demonstrated efficacy across a wide range of randomized controlled trials in children up to and older than 12 years of age. This work and the majority of efficacious PWMI have been based in large urban areas delivered through a hospital or medical center and the most recent childhood obesity treatment recommendations do not address geographically underserved audiences or settings where all members of an interdisciplinary team may not exist. As a result, there is no information on the degree to which evidence-based PWMIs have been translated into micropolitan (cities<50,000) and rural settings. This is an important issue when considering the prevalence of obesity is higher, socioeconomic status and access to preventive healthcare is lower, and 20% of the nation's populations reside in rural areas based on the most recent census data. A related issue is the potential mismatch between the resources and expertise used to deliver research and hospital-based PWMIs in urban, when compared to micropolitan and rural, areas. Thus, adoption, implementation, and sustainability may be limited in micropolitan and surrounding rural areas unless adaptations are made that leverage multiple systems within the community that interact with families and children and strategies include a balanced focus on reach and effectiveness to increase the likelihood of having a public health impact. To address these issues the research team has implemented an adapted version of the TLD in Kearney, Nebraska, developed and used training approaches for PWMI for underserved micropolitan settings, and conducted a number of implementation trials focused on planning for, and evaluating, PWMI reach, effectiveness, adoption, implementation and maintenance (RE-AIM). This includes research examining models of participant identification and engagement within settings where a large proportion of children are screened for obesity-schools and primary care pediatric clinics. Building Healthy Families (BHF), the investigators' TLD adaptation, includes the required or more contact hours through regular and frequent in-person contact with families and leverages the expertise and time of health professionals from a variety of local organizations. BHF has been implemented locally and successfully achieved clinically and statistically significant reductions in child BMI z-score (-0.27±0.22). Through collaborative efforts the research team has developed online resources for organizations interested in delivering PWMIs, training modules for related interventions, and participant-facing program materials that could be combined into a 'turn-key' approach for communities interested in reducing childhood obesity. The investigators preliminary work demonstrates that the adapted TLD intervention can achieve a similar magnitude of effect relative to previous efficacy trials, that the associated training materials and approaches can result in a high level of implementation fidelity, and that ongoing program adaptations to address local needs can be made. To date, the research team has not combined all of these approaches and materials as a turn-key package that could be adopted, adapted, and sustained in other micropolitan/rural communities.

The first aim is to collaboratively refine and develop an intervention package for the TLD that includes all of the materials necessary for others to implement the intervention in new micropolitan and rural locations. The second aim is to perform a rigorous, mixed-methods pilot implementation research study using an innovative community application process to identify 4 to 8 new communities to pilot test the utility of the packaged PWMI and training materials when coupled with a learning collaborative facilitation strategy and sustainability action planning process in supporting PWMI adoption, implementation, and sustainability when compared to receiving access to the packaged program and training materials alone. Additional outcomes will include start-up and ongoing costs while tracking intervention reach, representativeness, and effectiveness in reducing and maintaining child weight status relative to a matched cohort. The third aim is to use the pilot evaluation data and results of the sustainability action plan to refine program and training materials and develop a dissemination plan to move the program to other communities.

To complete these aims the investigators will engage an existing partnerships that includes local schools and pediatricians in Kearney, NE and the Great Plains IDeA Clinical and Translational Research Network Community Advisory Board who has identified childhood obesity treatment, particularly in rural areas, across North Dakota, South Dakota, and Nebraska as a priority. As is recommended, the approach will use an implementation research explanatory process, and outcome model to test hypotheses related to implementation and sustainability, engaging community/clinical partners in the implementation and sustainability process, and evaluate outcomes at both the individual and organizational level. Specifically, the Promoting Action on Research Implementation in Health Services (PARIHS) Framework will be used as the explanatory model and the RE-AIM framework to track individual reach, representativeness, effectiveness and organizational cost, adoption, implementation, and sustainability.

ELIGIBILITY:
Inclusion Criteria:

* Child 6 to 12 years of age
* Child with BMI percentile at or above the 95th percentile
* parents and/or guardian of child who meets the inclusion criteria

Exclusion Criteria:

* Child with major cognitive or physical impairments
* Child or parents/guardians with a contraindication for physical activity
* Families participating in a concurrent pediatric weight management intervention

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Program Implementation | up to 12 weeks
  % of objectives met during intervention sessions

SECONDARY OUTCOMES:
Body Mass Index percentile ranking | Calculated four times, baseline, 3-months, 6-months and 12 months
  Using standardized calculation for degree of childhood obesity as a function of height, weight, age and gender
Reach | measured once at enrollment
  number of children enrolled
Height in Meters | Measured once at baseline
  Measured in adults using a standard stadiometer
Weight in Kilograms | Measured 4 times; baseline, 3 months, 6-months and 12 months.
  Measured in adults using a research grade scale
Body Mass Index | Calculated 4 times; baseline, 3-months, 6-months and 12 months
  Calculated for adults from height and weight.
Community Adoption | 1 time at 3 months
  Number of communities and community organizations that respond to a call for applications
Cohort Adoption | up to 24 months
  The number of cohorts initiated in each community

OTHER OUTCOMES:
Cost | up to 24 months
  Cost of program adoption and implementation for communities will be tracked over the study using time tracking software to capture time spent on program activities for implementation staff.

CONTACTS AND LOCATIONS:
Overall Officials: Jennie Hill, PhD, Principal Investigator — University of Nebraska; Kate Heelan, PhD, Principal Investigator — University of Nebraska at Kearney

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data collected during the trial after deidentification.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available Jan 1, 2026 upon request.
Access Criteria: proposals should be sent to bhf@nebraska.edu. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Michaud TL, Hill JL, Heelan KA, Bartee RT, Abbey BM, Malmkar A, Masker J, Golden C, Porter G, Glasgow RE, Estabrooks PA. Understanding implementation costs of a pediatric weight management intervention: an economic evaluation protocol. Implement Sci Commun. 2022 Apr 5;3(1):37. doi: 10.1186/s43058-022-00287-1. PMID 35382891
- [Derived] Hill JL, Heelan KA, Bartee RT, Wichman C, Michaud T, Abbey BM, Porter G, Golden C, Estabrooks PA. A Type III Hybrid Effectiveness-Implementation Pilot Trial Testing Dissemination and Implementation Strategies for a Pediatric Weight Management Intervention: The Nebraska Childhood Obesity Research Demonstration Project. Child Obes. 2021 Sep;17(S1):S70-S78. doi: 10.1089/chi.2021.0170. PMID 34569848